CLINICAL TRIAL: NCT02250963
Title: Prognostic Accuracy of Coronary CT and Dobutamine Stress Echocardiography in Patient Undergoing Non-cardiac Surgery
Status: Terminated | Type: Observational
Sponsor: Gyeongsang National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GNUH-PANDA-01
Record Dates: First submitted 2014-09-15; First posted 2014-09-26 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Cardiac Complications of Care (& [Post Operative])
Keywords: Dobutamine Stress Echocardiography; Computed tomography coronary angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- DSE: Patients, who underwent Dobutamine Stress Echocardiography (DSE)
- CTCA: Computed tomography coronary angiography is going to perform with a 64-slice system (Brilliance 64, Philips Healthcare, Best, the Netherlands).

SUMMARY:
This study aimed to compare dobutamine stress echocardiography (DES) with computed tomography coronary angiography (CTCA) in patients with undergoing intermediate to high risk noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Elective surgery
2. Intermediate or high-risk noncardiac surgeries 1) intermediate risk surgery: intrathoracic, intraperitoneal, orthopedic,head and neck, and prostate 2) high risk surgery: vascular
3. Revised cardiac risk index score ≥1 (more than one of the following criteria) 1) vascular surgery, intraperitoneal, intrathoracic surgery 2) history of ischemic heart disease 3) history of heart failure 4) history of cerebrovascular disease 5) diabetes with insulin treatment 6) chronic kidney disease (serum creatinine > 2.0 mg/dL)

Exclusion Criteria:

1. Need for emergency surgery
2. Active cardiac conditions 1) recent (within 1 month) myocardial infarction 2) acute decompensated heart failure 3) severe valvular disease 4) fatal cardiac arrhythmia 5) acute pulmonary embolism 6) acute myocarditis
3. Relative contraindications or immeasurable coronary stenosis of the CTCA

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-cardiac surgery patients
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of DES vs. CTCA in the prediction of the postoperative hard cardiac events in patients undergoing intermediate to high risk noncardiac surgeries | 1 month
  Diagnostic performance includes sensitivity, specificity, positive and negative predictive values, and receiver operator curve area under the curve.
  Postoperative hard cardiac events were defined as cardiac death, non-fatal myocardial infarction.

SECONDARY OUTCOMES:
Diagnostic accuracy of DES vs. CTCA in the prediction of the perioperative all cardiovascular events in patients undergoing intermediate to high risk noncardiac surgeries. | 1 month
  Perioperative all cardiovascular events were defined as cardiac death, non-fatal myocardial infarction, pulmonary edema, ventricular fibrillation, new onset atrial fibrillation with hemodynamic compromise, complete heart block, pulmonary embolism, and prophylactic revascularization.
Diagnostic accuracy of DES and/or CTCA compared to revised cardiac risk score (RCRI) alone. | 1 month
  Incremental diagnostic accuracy changes with DES and/or CTCA compared to RCRI alone.
  Incremental diagnostic accuracy includes the area under the curve comparison analysis, integrated discrimination improvement, and net reclassification improvement.

OTHER OUTCOMES:
Diagnostic accuracy of blood viscosity test in the prediction of the perioperative cardiovascular events in patients undergoing intermediate to high risk noncardiac surgeries. | 1 month
  preoperative blood viscosity test using BVD (blood viscosity dynamic) system

CONTACTS AND LOCATIONS:
Locations (1):
- Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do, South Korea

REFERENCES:
- [Background] Ahn JH, Park JR, Min JH, Sohn JT, Hwang SJ, Park Y, Koh JS, Jeong YH, Kwak CH, Hwang JY. Risk stratification using computed tomography coronary angiography in patients undergoing intermediate-risk noncardiac surgery. J Am Coll Cardiol. 2013 Feb 12;61(6):661-8. doi: 10.1016/j.jacc.2012.09.060. PMID 23391198
- [Background] American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines; American Society of Echocardiography; American Society of Nuclear Cardiology; Heart Rhythm Society; Society of Cardiovascular Anesthesiologists; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine; Society for Vascular Surgery; Fleisher LA, Beckman JA, Brown KA, Calkins H, Chaikof EL, Fleischmann KE, Freeman WK, Froehlich JB, Kasper EK, Kersten JR, Riegel B, Robb JF. 2009 ACCF/AHA focused update on perioperative beta blockade incorporated into the ACC/AHA 2007 guidelines on perioperative cardiovascular evaluation and care for noncardiac surgery. J Am Coll Cardiol. 2009 Nov 24;54(22):e13-e118. doi: 10.1016/j.jacc.2009.07.010. No abstract available. PMID 19926002
- [Background] Das MK, Pellikka PA, Mahoney DW, Roger VL, Oh JK, McCully RB, Seward JB. Assessment of cardiac risk before nonvascular surgery: dobutamine stress echocardiography in 530 patients. J Am Coll Cardiol. 2000 May;35(6):1647-53. doi: 10.1016/s0735-1097(00)00586-6. PMID 10807472
- [Background] Labib SB, Goldstein M, Kinnunen PM, Schick EC. Cardiac events in patients with negative maximal versus negative submaximal dobutamine echocardiograms undergoing noncardiac surgery: importance of resting wall motion abnormalities. J Am Coll Cardiol. 2004 Jul 7;44(1):82-7. doi: 10.1016/j.jacc.2004.03.049. PMID 15234412
- [Derived] Ahn JH, Jeong YH, Park Y, Kwak CH, Jang JY, Hwang JY, Hwang SJ, Koh JS, Kim KH, Kang MG, Park JR. Head-to-head comparison of prognostic accuracy in patients undergoing noncardiac surgery of dobutamine stress echocardiography versus computed tomography coronary angiography (PANDA trial): A prospective observational study. J Cardiovasc Comput Tomogr. 2020 Nov-Dec;14(6):471-477. doi: 10.1016/j.jcct.2020.02.001. Epub 2020 Feb 4. PMID 32057706